CLINICAL TRIAL: NCT03978299
Title: Study of the Adequacy of the Requests of Prostate-Specific Antigen (PSA), Factors Associated With the False Negative and Positive Results and the Impact on Patient's Health
Brief Title: Factors Associated With PSA False Negative and False Positive Results and the Impact on Patient's Health.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital Universitario San Juan de Alicante (Other); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Blanca Juana Lumbreras Lacarra, Professor of Preventive Medicine and Public Health, Universidad Miguel Hernandez de Elche
Other Study IDs: PI17/01883.2; PI17/01883 (Other Grant/Funding Number: MINECO-FEDER)
Record Dates: First submitted 2019-05-28; First posted 2019-06-07 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Prostate-Specific Antigen /Blood
Keywords: Prostatic Neoplasms; False Positive Reactions; False Negative Reactions; Disease Management
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Positive PSA result: Men with a positive PSA test defined as:
  * Serum total PSA concentration is over 10 ng/ml.
  * Serum total PSA between 4 and 10 ng/ml if the value of the free PSA/total PSA fraction is under 25%, in at least in two determinations.
  Interventions: Diagnostic Test: Positive Prostate-Specific Antigen test result
- Negative PSA result: Men with a negative PSA test defined as:
  * Serum total PSA concentration is under 10 ng/ml.
  * Serum total PSA between 4 and 10 ng/ml if the value of the free PSA/total PSA fraction is over 25%.

INTERVENTIONS:
Diagnostic Test: Positive Prostate-Specific Antigen test result — Positive PSA test result as part of opportunistic screening or due to the presence of symptoms suggestive of disease.
  Groups: Positive PSA result

SUMMARY:
Objectives:

The primary aim of this study is to evaluate the outcomes of the determination of PSA for the early detection of prostate cancer or in the presence of symptoms, in general practice in two health departments of the Valencian Community (Spain).

Specific objectives:

1. To analyse the clinical and analytical factors associated with the presence of false positive and false negative results in PSA determinations in patients within the setting of opportunistic screening and in those with symptoms.
2. To evaluate the patient's clinical outcome, diagnostic and/or clinical and/or therapeutic interventions implemented in each patient according to the PSA value and the patient's clinical variables during the two years of follow-up. Furthermore, the investigadors will study whether this management is appropriate to the recommendations of the European Society of Urology.

DETAILED DESCRIPTION:
Sample size and recruitment procedure:

The investigators will select a cohort of patients with positive PSA results and a cohort of patients with negative results in each centre, to be followed for two years.

According to a review by the American Cancer Society, a value of PSA of 4 ng/ml had an estimated sensitivity of 21% to detect any type of prostate cancer and a specificity of 91%. The investigators estimate a prevalence of prostate cancer in this population not lower than 5% (given that the investigators include asymptomatic and symptomatic patients), with a 95% margin of error and 2% precision, the investigators will need to include 457 patients with a negative PSA result and 865 PSA-positive patients. Taking into account a 20% possible loss during follow-up, the investigators will increase to 572 patients with a negative PSA result (286 per centre) and 1,081 patients with a positive PSA result (541 per centre) who will be selected consecutively from among those included in the cross-sectional study until the investigators reach the proposed sample size. The investigators will use the initial randomized list (which included determinations during the first 6 months of 2018) to select patients who meet both negative and positive PSA criteria and if it is necessary, the investigators will continue to review analyses until the sample size is achieved.

Data collection procedure:

The investigators will follow both cohorts (positive and negative PSA results) for two years by reviewing their medical records (every 3 months for patients with a positive PSA result and annually for patients with a negative result). The following variables will be recorded: sociodemographic and clinical characteristics (patient who has the PSA determination as part of opportunistic screening or due to the presence of symptoms suggestive of disease), other comorbidities, toxic habits, previous history of cancer, family history, present pharmacological treatment and setting.

The investigators will evaluate the presence of false positive and negative results according to the latest recommendations of the European Association of Urology (specific objective 1).

The interventions performed after PSA determination and until the follow-up deadline, and their adaptation to the latest available recommendations (specific objective 2) will be evaluated separately by at least two investigators.

Data analysis plan The analysis will be performed using the Stata IC 15 program.

* Specific objective 1. The investigators will calculate the proportion of false positive and false negative results for the diagnosis of PCa and the associated variables. In the case of false positive tests, the investigators will also describe the time from a positive PSA result until PCa is ruled out using mean, standard deviation or median and interquartile ranges for the total population and relevant subgroups.
* Specific objective 2. The investigators will assess the probability of having a diagnostic, surgical or therapeutic intervention according to variables using risk ratio (statistical precision as for specific objective 1). If necessary, the investigators will use log-binomial regression estimating prevalence ratios. the investigators will also evaluate the agreement between the interventions performed and the available guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a PSA determination result in a routine health examination from the Health Department 17 and 19, in the Valencian Community (Spain)

Exclusion Criteria:

* Patients who have been previously diagnosed with prostate cancer.
* Patients who are being followed for previous high PSA values.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men over 18 from the Health Department 17 and 19, in the Valencian Community (these include General University Hospital of Sant Joan d'Alacant and General University Hospital of Alicante, respectively). These are referral hospitals for all individuals living in their catchment areas and belong to the National Health Care System (the majority of the population in Spain uses the National Health System (NHS) as the main medical service (the publicly funded insurance scheme covers 98.5% of the Spanish population).
  The investigators have not established maximum age limit.
Sampling Method: Probability Sample
Enrollment: 2527 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a false-positive result in the determination of serum PSA levels. | 2 years since PSA determination
  False positive result of the PSA determination defined as follows:
  If the PSA test is positive (meaning, serum total PSA level is over 10 ng/ml or serum total PSA level between 4 and 10 ng/ml if the value of the free PSA/total PSA fraction is under 25%, in at least in two determinations) and the result of digital rectal examination and/or subsequent biopsy is negative.
Proportion of patients with a false-negative result in the determination of serum PSA levels | 2 years since PSA determination
  False negative result of the PSA determination defined as follows:
  If the serum PSA value is negative (meaning, serum total PSA level is under 10 ng/ml or serum total PSA between 4 and 10 ng/ml if the value of the free PSA/total PSA fraction is over 25%) and the patient is diagnosed with prostate cancer in the subsequent follow-up.
Frequency of patients with appropriate diagnostic interventions performed in those with a positive serum PSA value according to "EAU - ESTRO - ESUR - SIOG Guidelines on Prostate Cancer". | 2 years since PSA determination
  Appropriateness of diagnostic interventions is defined as strategies that satisfies or not satisfies EAU recommendations with regard to the following issues:
  * Recommendations for clinical diagnosis of prostate cancer.
  * Recommendations for repeat-biopsy imaging.
Frequency of prostate cancer patients with an appropriate treatment protocol according to "EAU - ESTRO - ESUR - SIOG Guidelines on Prostate Cancer". | 2 years since PSA determination
  Appropriate treatment protocol is defined according to the EAU recommendations with regard to the number and type of therapeutic interventions carried out after prostate cancer diagnosis.
  The following information will be considered:
  * Surgical treatments.
  * Radiotherapeutic treatments.
  * Active therapeutic options outside surgery and radiotherapy.
  Each patient will be classified as "Appropriate according to guideline", "more intensive than guideline" or "less intensive than guideline".

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - San Juan de Alicante Hospital, Sant Joan d'Alacant, Alicante
  - FISABIO, Alicante

REFERENCES:
- [Background] Wolf AM, Wender RC, Etzioni RB, Thompson IM, D'Amico AV, Volk RJ, Brooks DD, Dash C, Guessous I, Andrews K, DeSantis C, Smith RA; American Cancer Society Prostate Cancer Advisory Committee. American Cancer Society guideline for the early detection of prostate cancer: update 2010. CA Cancer J Clin. 2010 Mar-Apr;60(2):70-98. doi: 10.3322/caac.20066. Epub 2010 Mar 3. PMID 20200110
- [Background] Chun FK, Epstein JI, Ficarra V, Freedland SJ, Montironi R, Montorsi F, Shariat SF, Schroder FH, Scattoni V. Optimizing performance and interpretation of prostate biopsy: a critical analysis of the literature. Eur Urol. 2010 Dec;58(6):851-64. doi: 10.1016/j.eururo.2010.08.041. Epub 2010 Sep 4. PMID 20884114
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Derived] Bernal-Soriano MC, Parker LA, Lopez-Garrigos M, Hernandez-Aguado I, Caballero-Romeu JP, Gomez-Perez L, Alfayate-Guerra R, Pastor-Valero M, Garcia N, Lumbreras B. Factors associated with false negative and false positive results of prostate-specific antigen (PSA) and the impact on patient health: Cohort study protocol. Medicine (Baltimore). 2019 Oct;98(40):e17451. doi: 10.1097/MD.0000000000017451. PMID 31577771